CLINICAL TRIAL: NCT05641961
Title: Utilizing a Mobile App to Help Survivors of Childhood Cancer Navigate Long-Term Follow-Up Care
Brief Title: Mobile App to Help Survivors of Childhood Cancer Navigate Long-Term Follow-Up Care
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Swim Across America (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 220813; NCI-2022-09452 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2022-11-29; First posted 2022-12-08 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Childhood Cancer; Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm
MeSH Terms: conditions — Neoplasms; Hematologic Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Survivorship Mobile Application (Experimental): Participants are seen in the survivorship clinic and receive education about potential late effects and the survivorship application on study. Participants enrolled in this study will be asked to complete two self-administered questionnaires at 4 time points. Questionnaires will be designed and made available electronically, to be completed on the participant's personal mobile device (e.g., mobile phone).
  Interventions: Behavioral: Survivorship mobile application; Other: Questionnaires

INTERVENTIONS:
Behavioral: Survivorship mobile application — Mobile phone application
  Other Names: Survivorship App
Other: Questionnaires — Questionnaires assessing cancer knowledge and system usability will be delivered to participants via Survivorship App

SUMMARY:
This clinical trial studies the effectiveness of a newly developed survivorship mobile application (app) designed for survivors, or their caregivers, of childhood cancer to help them better navigate long-term follow-up care. The survivorship app provides survivors access to their treatment history and follow-up recommendations, improves knowledge of their diagnosis, treatment, risks, and recommended follow-up care by using a message notification. The ability to quickly connect and establish care planning may enhance adherence to recommended follow-up.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the difference in survivor/caregiver knowledge and understanding of diagnosis, treatment information, and follow-up needs using the survivorship app.

SECONDARY OBJECTIVE:

I. To validate the usability and effectiveness of the survivorship mobile application.

OUTLINE:

Participants are seen in the survivorship clinic and receive education about potential late effects and the survivorship application on study. Participants then use the survivorship app for 4 months on study.

ELIGIBILITY:
Inclusion Criteria:

* Survivors of childhood cancer attending Survivorship Clinic at University of California, San Francisco (UCSF) OR caregivers of a childhood cancer survivor attending Survivorship Clinic at UCSF.
* Must have a mobile device (smartphone or smart-tablet) with service plan.
* Must have ability to read, write, and understand English language.

Exclusion Criteria:

* An individual who does not meet any of the criteria mentioned above will be excluded from participation in this study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-11-29 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in knowledge questionnaire score | Up to 4 months
  The knowledge of the participant will be measured using a 12-item questionnaire that assesses the awareness of their treatment and health issues in four categories: (1) diagnosis, (2) treatment, (3) risks, and (4) recommended follow-up. A scoring system has been devised which will give a score to each questionnaire out of 100 possible points. The change in participants knowledge scores >=20 points from baseline will be reported.

SECONDARY OUTCOMES:
System usability scale (SUS) score > 68 | Up to 2 months
  System Usability Scale (SUS) consists of a 10-item survey with five response options from Strongly agree to Strongly disagree. The scoring of positive questions is done as follows: The user's score is reduced by one point. For example, if the user's score is 4 for question 5, then the outcome score will be 3. The scoring of negative questions is done as follows: The user's score is subtracted from 5. For example, if the user's score is 3 for question 4, then the new score will be 2. After all the scores are determined, the sum of the scores is multiplied by 2.5 to make the range between 0 and 100. Scores above 68 are considered above average. The proportion of participants with an acceptable usability score > 68 will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Goldsby, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No